CLINICAL TRIAL: NCT04736238
Title: Peking University People's Hospital
Brief Title: Clinical Study on the Treatment of Chronic Instability of the Lateral Ankle Joint by Repairing the Anterior Talofibular Ligament Under Total Arthroscopy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Peking University People's Hospital (Other)
Responsible Party: Principal Investigator, Hailin Xu, Associate Professor, Peking University People's Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ATFLMicro
Record Dates: First submitted 2021-01-27; First posted 2021-02-03 (Actual); Last update posted 2021-02-03 (Actual); Status verified 2021-02

CONDITIONS: Anterior Talofibular Ligament Injury; Ankle Sprains
MeSH Terms: conditions — Ankle Injuries | interventions — Arthroscopy

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Trial group (Experimental): The patients who receive arthroscopic surgery.
  Interventions: Procedure: Arthroscopy surgery
- Control group (Other): The patients who receive BrostrÖm surgery.
  Interventions: Procedure: BrostrÖm surgery

INTERVENTIONS:
Procedure: Arthroscopy surgery — The patient receives intraspinal anesthesia or general anesthesia under supine position. Establish an anteromedial channel at the inner side of the tibial anterior tibial tendon at the level of the tibiotalar joint, and establish an anterolateral channel at the lateral angle of the talus. Exploring and clearing the ankle joint and dealing with possible combined injuries, such as talar cartilage injury, ankle impingement, and loose ankle joints. Then observe the lateral sulcus through the anterior medial channel, clean the synovium in the lateral sulcus, and explore the anterior talofibular ligament. A double-line anchor was inserted into the fibula side stop of the anterior talofibular ligament through the anterolateral channel. The anterior talofibular ligament was sutured using an outside-in technique in the anterior inferior safety zone of the distal end of the fibula. Fix the ankle joint with the suture after the dorsiflexion, neutral valgus position.
  Arms: Trial group
Procedure: BrostrÖm surgery — The patient receives intraspinal anesthesia or general anesthesia under supine position. The first ankle arthroscopy is performed to deal with possible combined injuries, such as talar cartilage injury, ankle impingement, and loose ankle joints. Then, open surgery was performed, and an arc incision was made at the anterior edge of the lateral malleolus to the tip of the fibula. After separating the subcutaneous tissue, the anterolateral joint capsule and talofibular ligament are exposed. A double-line anchor was placed at the fibular side stop of the anterior talofibular ligament. Tighten and suture the anterior talofibular ligament, anterolateral joint capsule, and extensor support belt with an anchor band. Fix the ankle joint with the suture after the dorsiflexion, neutral valgus position.
  Arms: Control group

SUMMARY:
This study mainly evaluated the clinical effect of total arthroscopic repair of the anterior talofibular ligament in the treatment of chronic instability of the lateral ankle. For patients with chronic instability of the lateral ankle, a randomized controlled trial was used to compare the curative effect, operation time, surgical complications, postoperative recurrence rate, postoperative recovery time and patients' satisfaction of the total arthroscopic repair of the anterior talofibular ligament surgery and the modified BrostrÖm surgery.

ELIGIBILITY:
Inclusion Criteria:

1. A history of acute lateral ankle sprain.
2. The patient has chronic instability of the lateral ankle joint, including functional instability or mechanical instability; functional instability refers to the patient's subjective ankle joint looseness or instability; mechanical instability refers to the presence of the ankle joint History of repeated sprains, positive examination of the front drawer test or positive X-ray examination of the stress position (inversion stress, anterior axial stress).
3. The ankle MRI suggested the anterior talofibular ligament injury.
4. It is invalid after 3 months of formal conservative treatment.

Exclusion Criteria:

1. Co-infection.
2. There was a previous ankle fracture in the affected limb.
3. The affected limb has previously undergone foot and ankle surgery.
4. Ankle inverted arthritis or Charcot joint disease.
5. Suffer from mental illness.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 44 (Estimated)
Dates: Start 2018-03-06 (Actual); Primary Completion 2021-06-30 (Estimated); Study Completion 2021-08-21 (Estimated)

PRIMARY OUTCOMES:
AOFAS ankle-hindfoot score | At 12 months after surgery

SECONDARY OUTCOMES:
Visual Analog Scale for Pain | At 12 months after surgery
  The pain VAS is available in the public domain at no cost [Arthritis Rheum 2003; 49: S96-104.]. Graphic formats for the VAS may be obtained online: http://www.amda.com/tools/library/whitepapers/hospiceinltc/appendix-a.pdf.
SF-36 Quality of Life Scale | At 12 months after surgery
Complications | At 12 months after surgery
  Wound infection, recurrence of ankle instability, ankle arthritis, rupture of anterior talofibular ligament.

CONTACTS AND LOCATIONS:
Locations (1):
- Peking University People's Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: No